CLINICAL TRIAL: NCT04213326
Title: Detecting Cancers Earlier Through Elective Plasma-based CancerSEEK Testing - Ascertaining Serial Cancer Patients to Enable New Diagnostic
Brief Title: Detecting Cancers Earlier Through Elective Plasma-based CancerSEEK Testing
Acronym: ASCEND
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: HEOR 24
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Results first posted 2023-01-18 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Early Cancer Detection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will have 6 (10 mL) biological samples (blood) collected in Streck circulating free DNA (cfDNA) tubes with a needle no larger than 21G. Tubes will be filled completely and then immediately mixed by gentle inversion 8-10 times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer Cohort: Subjects interested in the cancer cohort, will sign an informed consent, complete an optional survey, and have 60mLs of blood draw by a licensed phlebotomist.
- Non-Cancer Cohort: Subjects interested in the non-cancer cohort, will sign an informed consent, complete an optional survey, and have 60mLs of blood draw by a licensed phlebotomist.

SUMMARY:
This is a prospective, observational study of 1,000 subjects with known or suspected cancer and 2,000 subjects with no known cancer.

Potential participants will be asked questions to confirm their eligibility by a nurse navigator, study staff member, or physician.

Informed consent will be carried out for eligible subjects in accordance with applicable federal regulations and International Council for Harmonisation (ICH)/Good Clinical Practice (GCP) guidelines.

Subjects will then complete a survey, and study staff will draw 60 mL of blood and measure the height and weight of the subject.

Where available, data from the medical records of the cancer subjects will reviewed and collected. In addition, non-cancer subjects will be requested to allow access to their medical records as an optional portion of their informed consent.

DETAILED DESCRIPTION:
This is a prospective, observational study of 1,000 subjects with known or suspected cancer confirmed through pathology reports and/or clinical/radiographic data and 2,000 subjects with no known cancer. De-identified blood samples and clinical data will be collected from subjects to validate a classification algorithm for a new version of the CancerSEEK assay.

Potential participants will be asked questions to confirm their eligibility by a nurse navigator, study staff member, or physician to document screening including date of upcoming therapy or surgery for cancer patients if one has been scheduled, before providing informed consent to participate in the study. Study procedures outside of the pre-screening for eligibility will not be performed prior to the subject providing consent. Informed consent will be carried out in accordance with applicable federal regulations and International Council for Harmonisation (ICH)/Good Clinical Practice (GCP) guidelines. Prior to signing the informed consent form (ICF), potential participants will confirm that they understand the study and that they have no questions about the study.

The ICF may be offered by paper or electronically with the option to also review a paper copy provided by the nurse navigator or study coordinator either face-to-face on a tablet or via email. Potential participants will be given a phone number to call with any study specific questions. Copies of all signed consent forms will be stored centrally in a secure environment, and signed consent forms will thereby be available for verification by Thrive or its designee at any time.

Once the subject completes the survey, study staff will complete the blood draw and collect height and weight data. For some participants, their contact information and unique study identifier (ID) will be sent securely to a third-party vendor who will contact the subject within 24 hours to schedule the blood draw and height and weight measurements at a location convenient to the subject.

For all subjects, study staff and the third-party vendor performing the blood collection will verify the following before performing the blood draw and height and weight measurements: participant identity and age against a form of identification, that consent to participate has been given, that the participants in the cancer arm are still treatment naïve, and that they do not have a fever that could be caused by an infection. The blood collection vendor will ensure all required data are captured and included with the blood sample, that the sample is collected and packaged according to laboratory manual specifications, and that the sample is shipped to the indicated processing lab with the required expediency. Following all study visits, study staff and third party vendor staff will complete a visit checklist confirming all of the study activities that occurred.

Subjects in the Cancer cohort will be identified via nurse navigation, study staff or oncology physicians in local offices. The nurse navigator or study staff will verify eligibility through chart review and pre-screen, approach the subject about the study opportunity, and present the informed consent form. For participants enrolling electronically, participants will be presented with a secured tablet device on which the subject will watch a brief video about the study, read the informed consent and provide electronic consent. Some participants may also have the option of having the video, informed consent and survey emailed to them. Upon consent and enrollment, subjects will be assigned a unique subject study ID, which will be used to track the subject, their data and their biospecimen throughout study operations. Consented subjects will then be directed to complete a survey via the tablet device, email or paper. Participants will be allowed to skip questions in the survey or select the answer option "prefer not to answer." Subject data will be tracked in real-time by central study staff to ensure desired tumor type diversification and communicate enrollment strategy changes to the nurse navigators and study staff.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or greater
* Ability to understand the nature of this study and give written informed consent

CANCER COHORT:

Either of the following:

* Histologic diagnosis of cancer with no prior systemic or definitive therapy (any stage, including, inclusive of is-situ carcinoma)

Or

* Subject with high suspicion of cancer through radiological and/or clinical assessment who are scheduled for resection or biopsy within 6 weeks of study blood collection and have not received prior systemic or definitive therapy.

NON-CANCER COHORT

* No prior history of cancer

Exclusion Criteria:

ALL PATIENTS

* Evidence of active febrile infection prior to blood draw.
* Women who are pregnant or breast-feeding.
* History of an allogeneic bone marrow, stem cell transplant, or solid organ transplant.
* Judgment by the Investigator or study staff of any other reason that would prohibit the inclusion of the subject in the study.

CANCER COHORT

* Subjects newly diagnosed with a hematologic malignancy, primary central nervous system tumor, prostate cancer, or skin cancer (including melanoma).
* History of, or currently receiving, systemic or definitive cancer treatment including curative surgical resection, chemotherapy, radiation therapy, immunotherapy, and hormone therapy.

NON-CANCER COHORT

• None

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 3000 total subjects 2000 healthy volunteers 1000 cancer volunteers
Sampling Method: Probability Sample
Enrollment: 6400 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dax Kurbegov, MD, Principal Investigator — Sarah Cannon
Locations (14):
- United States (14):
  - Sarah Cannon, Thousand Oaks, California
  - Sarah Cannon, Denver, Colorado
  - Sarah Cannon, Fort Walton Beach, Florida
  - Sarah Cannon, Ocala, Florida
  - Sarah Cannon, Pensacola, Florida
  - Sarah Cannon, Augusta, Georgia
  - Sarah Cannon, Macon, Georgia
  - Sarah Cannon, Savannah, Georgia
  - Sarah Cannon, Kansas City, Kansas
  - Sarah Cannon, Overland Park, Kansas
  - Sarah Cannon, Independence, Missouri
  - Sarah Cannon, Las Vegas, Nevada
  - Sarah Cannon, Nashville, Tennessee
  - Sarah Cannon, Richmond, Virginia

REFERENCES:
- [Derived] Post C, Braun TP, Etzioni R, Nabavizadeh N. Multicancer Early Detection Tests: An Overview of Early Results From Prospective Clinical Studies and Opportunities for Oncologists. JCO Oncol Pract. 2023 Dec;19(12):1111-1115. doi: 10.1200/OP.23.00260. Epub 2023 Oct 18. PMID 37851937

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cancer Cohort | Non-Cancer Cohort
Started | 937 | 5463
Completed | 727 | 3893
Not Completed | 210 | 1570
Not completed — Consent withdrawn | 51 | 241
Not completed — Lost to Follow-up | 50 | 902
Not completed — Protocol Violation | 3 | 25
Not completed — Participant eligibility changed | 106 | 19
Not completed — SCRI confirmed to be withdrawal | 0 | 16
Not completed — Incomplete study visit | 0 | 367

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cancer Cohort | Non-Cancer Cohort | Total
Number analyzed (Participants) | 727 | 3893 | 4620
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (9) | 62 (8) | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The numbers analyzed in the sex category differ from the overall participants due to missing data for 26 subjects. Sex was not able to be collected for 19 subjects in the cancer cohort and 7 in the non-cancer cohort.
  Participants
    number analyzed (Participants) | 708 | 3886 | 4594
    Female | 451 | 2374 | 2825
    Male | 257 | 1512 | 1769
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 525 | 3360 | 3885
  Race: Black | 83 | 316 | 399
  Race: Asian/Pacific Islander | 3 | 53 | 56
  Race: Native American/Alaskan | 1 | 14 | 15
  Race: Other | 11 | 65 | 76
  Race: Missing | 104 | 85 | 189
Region of Enrollment [Number; unit: participants]
  United States | 727 | 3893 | 4620

OUTCOME MEASURES:

1. Primary Outcome: Study Data and Samples Were Used for CancerSEEK Assay Development
Description: The primary objective of the study is to collect blood samples from known cancer and non cancer participants. These blood samples were used to calibrate the CancerSEEK assay. There was no pre-defined performance threshold.
Time Frame: 6 months
Population: Blood samples collected to be used to calibrate the CancerSEEK assay.
Measure: Count of Participants; unit: Participants
Arm/Group | Cancer Cohort | Non-Cancer Cohort
Number analyzed (Participants) | 727 | 3893
Participants
  Not withdrawn, With Blood Draw | 712 | 3870
  Withdrawn, With Blood Draw (lost to follow up) | 5 | 14
  Withdrawn after Blood Draw | 10 | 9

ADVERSE EVENTS:
Time Frame: Adverse Events collected at blood draw.
Arm/Group | Cancer Cohort | Non-Cancer Cohort
All-Cause Mortality (participants affected / at risk) | 0/727 | 0/3893
Serious Adverse Events (participants affected / at risk) | 0/727 | 0/3893
Other Adverse Events (participants affected / at risk) | 0/727 | 0/3893

LIMITATIONS AND CAVEATS:
With the acquisition of Thrive Earlier Detection by Exact Science in early 2021, the primary objective shifted. The study data and samples were used for CancerSEEK assay development only and no endpoint analysis was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT04213326/Prot_SAP_000.pdf